CLINICAL TRIAL: NCT03417713
Title: Clinical Evaluation of the OEC Elite MD for Vascular Procedures
Brief Title: Clinical Evaluation of the OEC Elite MD for Vascular Procedures at Hamilton General Hospital
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 104-2017-GES-0005
Record Dates: First submitted 2018-01-12; First posted 2018-01-31 (Actual); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-10

CONDITIONS: Interventional Vascular Conditions
MeSH Terms: interventions — Fluoroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All Subjects: This group/cohort is expected to be representative of the general population that would require mobile fluoroscopic imaging with C-arm devices, such as OEC Elite.
  Interventions: Device: Fluoroscopic imaging with the OEC Elite Device

INTERVENTIONS:
Device: Fluoroscopic imaging with the OEC Elite Device — Vascular, gastrointestinal (GI), urology or pain management procedures for which use of the OEC Elite system in the vascular configuration would be prescribed.

SUMMARY:
The purpose of this study is to collect feedback on imaging guidance adequacy from physicians who use the OEC™ Elite CFD Mobile Fluoroscopy System-Motorized Configuration to perform surgical procedures for which the use of mobile fluoroscopy is prescribed per standard of care.

Up to 40 eligible subjects will be enrolled and have their clinically indicated procedure completed using the investigational device.

Following completion of each subject's procedure, the investigators will complete a User Survey specific to the workflow and guidance adequacy of the OEC Elite device. The survey will consist of a series of questions on the use of the system as well as anonymized image data.

After all subjects' procedures are completed at a given site, the site investigator will review survey data from the study subjects enrolled at the site and document his/her assessment of the overall acceptability of the system for use in a clinical environment.

There is no statistical hypothesis being tested in this study. Results will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 85 years (≥18 and ≤85 years old);
2. Clinical indication for procedures including vascular, gastrointestinal (GI), urology or pain management for which mobile fluoroscopy has been prescribed for image guidance;
3. Able and willing to comply with study procedures; and
4. Able and willing to provide written informed consent to participate.

Exclusion Criteria:

1. Pregnant or suspected to be pregnant based on the opinion of and as documented by a medically qualified physician investigator;
2. Expected to be at increased risk due to study participation (e.g. due to allergies, sensitivities), in the medical opinion of an investigator; or
3. Previously participated in this study, or enrolled in another active GEHC study or other research study that could be expected to interfere with participation in study procedures, in the opinion of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults undergoing vascular, gastrointestinal (GI), urology or pain management procedures for which use of the OEC Elite system in the vascular configuration would be prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 33
Completed | 30
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: Years] | 69.9 [55 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Image Guidance Adequacy Collected Via Survey Questionnaire
Description: Number of participants whose procedures were completed using the investigational device.
Time Frame: Approximately 2 months (duration of subject enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Number of Investigator Procedure Surveys Assessed by Survey Questionnaire
Description: To collect image data acquired during clinical procedures and to collect investigator feedback via surveys on the use of the system during clinical procedures.
Time Frame: Approximately 2 months (duration of subject enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse events were collected from when the subject entered the study to when they completed study procedures
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=30)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03417713/Prot_SAP_000.pdf